CLINICAL TRIAL: NCT02658955
Title: Changing Technique of Abdominal Wall Closure According to European Hernia Society (EHS) Guidelines in a General Hospital
Brief Title: Changing Technique of Abdominal Wall Closure (PHACPA)
Acronym: PHACPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital del Mar (Other)
Responsible Party: Principal Investigator, José A. Pereira, MD, Hospital del Mar
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMar
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Closure of Abdominal Wall
Keywords: Abdominal wall closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Short stitch (Experimental): Patients in which abdominal wall is closed by short stitch technique
  Interventions: Procedure: Short stitch
- Large stitch (No Intervention): Patients who didn't receive properly closure according with the protocol

INTERVENTIONS:
Procedure: Short stitch — Surgeons will receive instructions to change the technique of abdominal wall closure
  Arms: Short stitch

SUMMARY:
Implementing guidelines of EHS for abdominal wall closure in all specialities of a General Hospital. Migrating from large stitch technique to short stitch technique.

DETAILED DESCRIPTION:
Surgeons will receive instruction about new techniques of closure of the abdomen and will practice in models and receive a certification previously to implement in their surgical practice the new technique.

Results will be monitorised and compared with previous cohort of patients. A protocol of closure will be implemented. Patients without risk factors will receive a laparotomy closure with "short stitch" technique and patients with risk factor for developing incisional hernia or burst abdomen and aditional profilactic suprafascial mesh.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated on by laparotomy

Exclusion Criteria:

* Previous mesh
* Concomitant hernia repair

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1164 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Incisional hernia and burst abdomen rate | One year
  Analysis of the number of incisional hernia and burst abdomen after one year follow-up

SECONDARY OUTCOMES:
Rate of fulfillment of the protocol | One year
  Analysis of results related with the fulfillment of the protocol
Complication rate | One month
  Analysis of complications related with the closure technique
Mesh complications rate | One year
  Analysis of mesh related complications in patients with a prophylactic mesh

CONTACTS AND LOCATIONS:
Overall Officials: José A. Pereira, MD, Principal Investigator — Surgeon
Locations (1):
- José A. Pereira, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No